CLINICAL TRIAL: NCT01207024
Title: Assessment of Knee Arthrosis in Severely Obese Patients After Bariatric Surgery.
Brief Title: Assessment of Knee Arthrosis After Bariatric Surgery
Acronym: BASIK
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P071225
Record Dates: First submitted 2010-08-26; First posted 2010-09-22 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Bariatric Surgery Candidate
Keywords: knee arthrosis; obesity; MRI; bariatric surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- knee MRI: knee MRI for all patients undergoing bariatric surgery as usual care
  Interventions: Other: knee MRI

INTERVENTIONS:
Other: knee MRI — knee MRI before surgery (inclusion) and one year after

SUMMARY:
Impact of loss of weight on knee arthrosis has not been thoroughly studied. The primary goal of this study is to compare the MRI parameters (aspect of cartilage and oedema of spongious sub-chondral bone) before and one year after bariatric surgery.

Knee MRI is not currently part of the investigations preceding bariatric surgery.

DETAILED DESCRIPTION:
Assessment of knee arthrosis in severely obese patients after bariatric surgery.

Impact of loss of weight on knee arthrosis has not been thoroughly studied. The primary goal of this study is to compare the MRI parameters (aspect of cartilage and oedema of spongious sub-chondral bone) before and one year after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* bariatric surgery
* IMC >= 35

Exclusion Criteria:

* those of bariatric surgery
* contra-indication to MRI
* pregnancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inclusion Criteria:
  * bariatric surgery
  * IMC >= 35
  Exclusion Criteria:
  * those of bariatric surgery
  * contra-indication to MRI
  * pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-02; Primary Completion 2013-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
variation of knee joint space thickness | 24 hours, one year
  Joint space variation in percentages (mean joint space variation calculated for each patient group). Mean joint space comparison between 2 groups of obese patients: patients with Bypass surgery versus patients without surgery.
proportion of patients with pain | 1 year
  proportion of patients with Pain Scores on the Visual Analog Scale ≥ 30/100 (for at least one knee). Comparison at one year after bariatric surgery versus inclusion.

SECONDARY OUTCOMES:
prevalence of atherosis | 24 hours
  Pain Scores on the Visual Analog Scale >= 3 and/or radiological signs of atherosis
mean pain and disability | 24 hours
  mean Pain Scores on the Visual Analog Scale and mean value of KOOS index for knee function.
evolution of KOOS score after surgery | 6 months, 1 year and two years
  Among the 80 patients undergoing surgery, comparison of KOOS function score before surgery versus 6 months, 1 year and two years after surgery.
evolution of pain scores after surgery | 6 months, 1 year, 2 years
  Among the 80 patients undergoing surgery, comparison of mean Pain Scores on the Visual Analog Scale before surgery versus 6 months, 1 year and two years after surgery.
evolution of the proportion of patients in pain | 6 months, 1 year and two years
  Among the 80 patients undergoing surgery, comparison of the proportion of patients with Pain Scores on the Visual Analog Scale ≥ 30/100 before surgery versus 6 months, 1 year and two years after surgery.
evolution of knee MRI parameters after surgery | 6 months, 1 year and two years
  Among the 80 patients undergoing surgery, comparison of the MRI parameters (T2, cartilage volume, œdema of sub-chondral spongious bone) before surgery versus 6 months, 1 year and two years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Dion, MD, Phd, Principal Investigator — Louis Mourier University Hospital (AP-HP)
Locations (1):
- Louis Mourier hospital (AP-HP), Colombes, France